CLINICAL TRIAL: NCT07309263
Title: Comparing the Effects of Smart App-Assited Super-Slow Jogging and Stationary Cycling on Respiratory Function and Aerobic Fitness in College Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fooyin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 114-0561; 114-2813-C-242-003-B (Other Grant/Funding Number: National Science and Technology Council, Taiwan)
Record Dates: First submitted 2025-11-21; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-08

CONDITIONS: Sedentary Lifestlye; Young Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Super slow jogging (Experimental): A smart app will provide pacing assistance, adjusting step frequency weekly: Week 1: 150 steps per minute Week 2: 180 steps per minute Week 3: 190 steps per minute Week 4: 200 steps per minute
  Interventions: Behavioral: Super slow jogging
- moderate exercise training (Experimental): Continuous cycling training at moderate intensity of 60% VO₂max
  Interventions: Behavioral: moderate exercise training
- Control (Placebo Comparator): not perform any exercise training
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Super slow jogging — This study is a randomized controlled trial employing simple randomization, where participants draw lots to assign groups. The experiment comprises three groups: the super-slow jogging group, the stationary bicycle group, and the control group. Both exercise intervention groups underwent 50-minute training sessions comprising a 10-minute warm-up, 30-minute main exercise, and 10-minute cool-down.
  Super-Slow Jogging Group: Utilized a smart app for pacing assistance, adjusting step frequency weekly:
  Week 1: 150 steps/minute Week 2: 180 steps/minute Week 3: 190 steps/minute Week 4: 200 steps/minute Stationary Cycling Group: Participants will engage in continuous cycling training at moderate intensity (60% VO₂max).
  Control Group: No exercise training intervention.
  Arms: Super slow jogging
Behavioral: moderate exercise training — This study is a randomized controlled trial employing simple randomization, where participants draw lots to assign groups. The experiment comprises three groups: the super-slow jogging group, the stationary bicycle group, and the control group. Both exercise intervention groups underwent 50-minute training sessions comprising a 10-minute warm-up, 30-minute main exercise, and 10-minute cool-down.
  Super-Slow Jogging Group: Utilized a smart app for pacing assistance, adjusting step frequency weekly:
  Week 1: 150 steps/minute Week 2: 180 steps/minute Week 3: 190 steps/minute Week 4: 200 steps/minute Stationary Cycling Group: Participants will engage in continuous cycling training at moderate intensity (60% VO₂max).
  Control Group: No exercise training intervention.
  Arms: moderate exercise training
Behavioral: Control — This study is a randomized controlled trial employing simple randomization, where participants draw lots to assign groups. The experiment comprises three groups: the super-slow jogging group, the stationary bicycle group, and the control group. Both exercise intervention groups underwent 50-minute training sessions comprising a 10-minute warm-up, 30-minute main exercise, and 10-minute cool-down.
  Super-Slow Jogging Group: Utilized a smart app for pacing assistance, adjusting step frequency weekly:
  Week 1: 150 steps/minute Week 2: 180 steps/minute Week 3: 190 steps/minute Week 4: 200 steps/minute Stationary Cycling Group: Participants will engage in continuous cycling training at moderate intensity (60% VO₂max).
  Control Group: No exercise training intervention.
  Arms: Control

SUMMARY:
As health awareness continues to rise, more people are prioritizing exercise to improve physical condition and enhance overall fitness. For those lacking exercise habits, selecting a simple, accessible, and effective workout becomes crucial. Against a backdrop of prolonged sitting and inactivity, "super slow jogging" is gaining attention. This aerobic exercise involves a slow walking pace and low intensity, yet burns more calories than regular walking, making it an ideal entry-level activity for beginners or those with lower fitness levels. This study aims to investigate whether incorporating super slow jogging training can effectively enhance cardiorespiratory fitness and respiratory function, comparing its outcomes with other exercise types. The purpose of this experiment is academic research, primarily exploring the impact of exercise intervention on physiological functions. It is not intended for health screening or medical diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* required no regular exercise training in the past six months
* ability to safely perform high-intensity cycling exercise

Exclusion Criteria:

* musculoskeletal limitations that prevented cycling exercise
* recent infection
* known cardiopulmonary disease or medical history affecting cardiovascular or respiratory function
* smoking
* use of medications that may influence cardiopulmonary responses to exercise
* other contraindications to exercise testing according to the American College of Sports Medicine (ACSM) guidelines

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Cardiopulmonary Fitness | Before intervention and the end of intervention at 12 weeks
  VO2max (ml/kg/mL)
Baseline anthropometric of the participants | Before intervention and the end of intervention at 12 weeks
  Age (yr)
Cardiopulmonary Fitness | Before intervention and the end of intervention at 12 weeks
  VEmax (L/min)
Cardiopulmonary Fitness | Before intervention and the end of intervention at 12 weeks
  AT% (%VO₂max)
Cardiopulmonary Fitness | Before intervention and the end of intervention at 12 weeks
  Resting O₂ pulse (mL·beat-¹)
Cardiopulmonary Fitness | Before intervention and the end of intervention at 12 weeks
  Max O₂ pulse (mL·beat-¹)
Cardiopulmonary Fitness | Before intervention and the end of intervention at 12 weeks
  MIP (cmH2O)
Cardiopulmonary Fitness | Before intervention and the end of intervention at 12 weeks
  MEP (cmH2O)
Baseline anthropometric of the participants | Before intervention and the end of intervention at 12 weeks
  Height (cm)
Baseline anthropometric of the participants | Before intervention and the end of intervention at 12 weeks
  Weight (kg)
Baseline anthropometric of the participants | Before intervention and the end of intervention at 12 weeks
  BMI (kg/m²)

SECONDARY OUTCOMES:
Lung function | Before intervention and the end of intervention at 12 weeks
  FEV1 (L)
Lung function | Before intervention and the end of intervention at 12 weeks
  FVC (L)
Lung function | Before intervention and the end of intervention at 12 weeks
  FEV₁/FVC (%)
Lung function | Before intervention and the end of intervention at 12 weeks
  FEF25-75% (L·s-¹)
Lung function | Before intervention and the end of intervention at 12 weeks
  PEF (L·min-¹)
Lung function | Before intervention and the end of intervention at 12 weeks
  MVV (L·min-¹)
Lung function | Before intervention and the end of intervention at 12 weeks
  Breathing reserve (%)
Lung function | Before intervention and the end of intervention at 12 weeks
  Dynamic Index (DI%)

CONTACTS AND LOCATIONS:
Locations (1):
- No. 151, Jinxue Rd., Kaohsiung City, Daliao, Taiwan

IPD SHARING:
Plan to Share IPD: No